CLINICAL TRIAL: NCT02753010
Title: Gastric Emptying Time of a Carbohydrate-rich Drink in Elderly Patients With Acute Hip Fracture: a Pilot Study
Brief Title: Gastric Emptying in Elderly With Hip Fracture
Acronym: GASEMPHIP
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Hellström, Professor, MD, PhD, Uppsala University
Other Study IDs: GASEMPHIP
Record Dates: First submitted 2016-04-17; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Gastroparesis; Hip Fracture; Mild Insufficient Nutrition
MeSH Terms: conditions — Gastroparesis; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acute hip fracture: Women preoperatively with acute hip fracture with gastric emptying of carbohydrate-rich beverage
  Interventions: Procedure: Gastric emptying of carbohydrate-rich beverage
- Elective hip replacement: Women on waiting list for elective hip replacement with gastric emptying of carbohydrate-rich beverage
  Interventions: Procedure: Gastric emptying of carbohydrate-rich beverage
- Healthy volunteers: Healthy female volunteers with gastric emptying of carbohydrate-rich beverage
  Interventions: Procedure: Gastric emptying of carbohydrate-rich beverage

INTERVENTIONS:
Procedure: Gastric emptying of carbohydrate-rich beverage — Old women with acute hip fracture with intake of carbohydrate-rich beverage in order to improve metabolic control. Gastric emptying studied for retention in the elderly with acute trauma.
  Other Names: Gastric emptying of beverage (Nutricia Preop; Numico)
  Groups: Acute hip fracture
Procedure: Gastric emptying of carbohydrate-rich beverage — Old women on waiting list for hip joint replacement with intake of carbohydrate-rich beverage in order to improve metabolic control. Gastric emptying studied as comparator in the elderly without acute trauma..
  Other Names: Gastric emptying of beverage (Nutricia Preop; Numico)
  Groups: Elective hip replacement
Procedure: Gastric emptying of carbohydrate-rich beverage — Young healthy women with intake of carbohydrate-rich beverage in order to improve metabolic control. Gastric emptying studied as comparator in young women.
  Other Names: Gastric emptying of beverage (Nutricia Preop; Numico)
  Groups: Healthy volunteers

SUMMARY:
The gastric emptying of 400 ml 12.6% carbohydrate rich drink is investigated in elderly women, age 75-100, with acute hip fracture. The emptying time will be assessed by the paracetamol absorption technique, and lag phase and gastric half-emptying time compared with two gender-matched reference groups: elective hip replacement patients, age 45-71, and healthy volunteers, age 28-55.

DETAILED DESCRIPTION:
Patients with hip fracture are submitted to prolonged fasting before surgery is undertaken. This is deleterious for their metabolic condition and slows recovery after surgery.

A carbohydrate-rich beverage is taken immediately before surgery and gastric emptying rate is assessed in elderly (75-100 yo) women prior to surgery for acute hip fracture. As comparator another two groups of women are used; one scheduled for elective surgery for hip replacement due to osteoarthritis; another healthy female volunteers.

On the day of surgery the primary study group of acute hip fracture is given a carbohydrate-rich beverage 400 ml, total 200 kcal in combination with paracetamol 1.5 g. Blood samples are intermittently drawn during 180 minutes to measure recovery of paracetamol in plasma and gastric emptying rate calculated according to previously published principles. In the same manner a group of women on waiting list for hip replacement surgery due to osteoarthritis are enrolled for estimation of gastric emptying rate. In addition, another group of completely healthy women are enrolled for assessment of gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* female gender, age 75 years or above, and hip fracture within 24 hours of admission.

Exclusion Criteria:

* gastro-esophageal reflux disease, peptic ulcer disease, gastrointestinal motility disorder, pulmonary or cardiac disease, pharmacological treatment with motility-stimulating agents such as dopamine-receptor blockers or macrolides, as well as previous long-term opioids or acid inhibitory agents, or cognitive impairment at the discretion of the investigator

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly women with acute hip fracture awaiting surgery within the next 24 hours. Since surgery is performed early next morning, patients will be kept fasted for prolonged periods of time with only continuous line of glucose 5% or 10% solution. This will not evoke any insulin response which is needed for controlled metabolic condition.
  In addition: Patients elective for hip replacement, healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | 0-180 minutes

SECONDARY OUTCOMES:
Gastric lag phase | 0-60 minutes
Pulmonary aspiration | 0-180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Hedström, MD, PhD, Study Director — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hellstrom PM, Samuelsson B, Al-Ani AN, Hedstrom M. Normal gastric emptying time of a carbohydrate-rich drink in elderly patients with acute hip fracture: a pilot study. BMC Anesthesiol. 2017 Feb 15;17(1):23. doi: 10.1186/s12871-016-0299-6. PMID 28202056